CLINICAL TRIAL: NCT06656754
Title: Error-enhanced Learning & Recovery in 2 & 3 Dimensions
Brief Title: R01.Aim 2.Study 1: IsoReach
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Lanphier Patton, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STU00220740
Record Dates: First submitted 2024-09-04; First posted 2024-10-24 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Reaching condition (Experimental): In this arm the participant participates in "Isometric Reaching" in which they are not allowed to freely reach to the target, instead the forces they apply on the robot handle drives a reaching arm simulation
  Interventions: Other: Isometric Reaching
- Control Reaching condition (No Intervention): In this condition the participant moves toward target freely and the visual feedback is based on hand position and not an arm simulation.

INTERVENTIONS:
Other: Isometric Reaching — The intervention of "Isometric Reaching" is the process of restricting the participant's hand movement in place, while using the forces they apply to the robot handle to drive a reaching arm simulation
  Arms: Isometric Reaching condition

SUMMARY:
To determine the effects of 3D isometric movement training in healthy participants and impaired participants due to a stroke.

DETAILED DESCRIPTION:
Researchers have found that neurotypical adults are able to train movement skills when sensory sources, such as proprioception, are altered using isometric conditions and visual feedback in a two-dimensional environment.Building off this knowledge, the investigators plan to apply similar techniques to both neurotypical adults and stroke survivors with impaired movement, but in a three-dimensional environment. The investigators will ask participants to practice a unilateral virtual reality targeted reaching task using a robotic arm in a 3D visual display system mounted over the arm. Participants will be given visual feedback of their arm through a virtual avatar displayed on the screen. First, they will complete unconstrained targeted reaching and then complete targeted reaching with the robotic arm constrained in a fixed position ("isometric" movement). The forces applied to constrain the robotic arm will be translated to the virtual avatar arm on the screen, and it will look as if their arm is moving. The investigators will compare perpendicular errors (maximum difference between the ideal reaching trajectory and the actual) made in unconstrained and constrained movement conditions. The investigators aim to determine if the two movement conditions yield similar error responses when sensory sources are altered in a 3D environment.

ELIGIBILITY:
Inclusion criteria, neurotypical participants

* 18 years old

No history of stroke

Ability to provide informed consent .

Exclusion criteria, neurotypical participants

Severe medical problems (including cardiovascular, orthopedic, or neurological)

Medical problems affecting movement, range of motion, strength, or coordination of the upper extremities.

Visual deficits that would influence the ability to perform the experiment . This will be assessed using the following assessments:

1. Visual field deficits will be assessed using the BIVABA acuity testing. (cutoff score > 20/100)
2. Depth perception deficits will be assessed using the Stereofly test (require at least an angle of stereopsis at 16 inches is 3,552 seconds of arc).

   4) Blood pressure above 140 systolic and/or 90 diastolic mmHG

   5) Blood oxygen reading of less than 92% by finger pulse oximeter testing.

   Inclusion Criteria , Stroke participants
   * 18 years old

   Chronic stroke (8+ months post)

   Available medical records and radiographic information about lesion locations

   Hemiparesis

   Primary motor cortex involvement

   Some degree of both shoulder and elbow movement capability

   Exclusion Criteria , Stroke participants

   Bilateral paresis

   Aphasia, cognitive impairment, or affective dysfunction that would influence the ability to perform the experiment, This will be assessed using the Mini Mental State Examination31, with cut-off scores (adjusted for education level) as follows:

   Participants whose education are 7th grade or lower, a score 22 or lower

   Participants whose education attainment level is 8th grade or some high school (but not a graduate), a score of 24 or lower

   Participants whose education attainment level is high school graduate, a score of 25 or lower

   Participants whose education attainment level is some college or higher, a score 26 or lower

   Visual deficits, and hemispatial neglect that would prevent the participants from seeing the targets. A vision test will be done if the participant indicates in their screen that their stroke has affected their vision. This will be tested using the following assessments:

   Visual field loss will be assessed using the BIVABA acuity test10. (cutoff score > 20/100)

   Visual Extinction and Inattention using Star Cancellation Test9. (cutoff score of <44)

   Depth perception deficits will be assessed using the Stereofly test (require at least an angle of stereopsis at 16 inches is 3,552 seconds of arc).

   Modified Ashworth score of 4 at shoulder or elbow joints.

   Rated below 15 on the FMUE scale

   Inability to provide an informed consent

   severe current medical problems

   Severe sensory deficit in the affected limb (Cannot be absent in any part of affected UE)

   diffuse/multiple lesion sites or multiple stroke events

   Inability to attain and maintain testing positions

   Botox or other botulinum toxin injection to the affected upper extremity within the previous 4 months

   Concurrent participation in upper extremity rehabilitation either as part of a research intervention protocol or a prescribed therapy

   Neurological, neuromuscular, or orthopedic diseases (i.e. injuries to your affected arm or hand)

   Other neurological issues (Parkinson's, CP)

   Blood Pressure above 140 systolic and/or 90 diastolic mmHg

   Blood oxygen reading of less than 92% on finger pulse oximetry testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Perpendicular Error | through study completion, an average of 1 year.
  Maximum distance between the ideal reaching trajectory and the actual trajectory made in unconstrained and constrained movement conditions

CONTACTS AND LOCATIONS:
Overall Officials: James L Patton, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States